CLINICAL TRIAL: NCT00801047
Title: Comparison of the Efficacy Intravenous Remifentanil PCA and Epidural PCEA for Labor Analgesia
Brief Title: Intravenous Remifentanil Patient-controlled Analgesia (PCA) and Epidural Patient Controlled Epidural Analgesia (PCEA) for Labor Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Carolyn Weiniger, Hadassah Medical Organization
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: rem-epi-nov-2008- HMO-CTIL
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2010-02

CONDITIONS: Labor; Pain
Keywords: Epidural; Labor; Remifentanil
MeSH Terms: conditions — Pain | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Epidural group
  Interventions: Drug: Bupivacaine epidural
- 2 (Active Comparator): Remifentanil iv PCA
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Bupivacaine epidural — Bupivacaine 0.1%, fentanyl 1 mic/kg
  Arms: 1
Drug: Remifentanil — 40-50 mic per 1-2 min via PCA
  Arms: 2

SUMMARY:
Women requesting analgesia do not always wish to receive a potent analgesic method, and may fear the risks of epidural analgesia.

Study Aim: To determine whether remifentanil is effective for labor analgesia when compared with standard treatment (epidural analgesia).

ELIGIBILITY:
Inclusion criteria:

* Healthy women
* American Society of Anesthesiologists physical status class I or II
* Body weight less than 110 kg
* In active labor (including induced labor and premature rupture of membranes)
* Cervical dilatation at 2-6 cm
* Regular contractions
* Age between 18 and 40 years old
* Gestational age greater than 36 completed weeks
* Singleton pregnancy and vertex presentation

Exclusion criteria:

* Contraindication for epidural analgesia (bleeding diathesis, neuropathy, severe scoliosis, previous spine surgery, local anesthetic allergy)
* Narcotic administration in the previous 2 hours
* Previous uterine surgery
* Pre-eclampsia and the inability to adequately understand the consent form
* Blocked nose, and any indication patient for whom epidural analgesia is medically indicated (cardiac disease, suspected difficult airway)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Primary analgesia end-point: VAS pain Score | 1-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn F Weiniger, MB ChB, Principal Investigator — Hadassah HMO
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Hill D. Remifentanil patient-controlled analgesia should be routinely available for use in labour. Int J Obstet Anesth. 2008 Oct;17(4):336-9. doi: 10.1016/j.ijoa.2008.03.005. No abstract available. PMID 18617388